CLINICAL TRIAL: NCT05665868
Title: The Construction and Empirical Study of Symptom Management and Integrated Care Strategy for Gastrointestinal Stromal Tumor Patients With Targeted Therapy Based on MRC Framework
Brief Title: Study on Integrated Nursing Strategy for Patients With Gastrointestinal Stromal Tumors After Targeted Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022-LCYJ-MS-30
Record Dates: First submitted 2022-11-27; First posted 2022-12-27 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-11

CONDITIONS: Nursing Caries; Gastrointestinal Stromal Tumors
MeSH Terms: conditions — Gastrointestinal Stromal Tumors

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group based on integrated care mode (Experimental): ① Obtain the health records of patients receiving targeted treatment of gastric stromal tumors in the big data platform; ② Patients upload health data, disease symptoms, complete questionnaires, health consultation and other functions; ③ The platform can regularly send audit reminders, automatically analyze the data uploaded and saved by patients, automatically and intelligently intervene when abnormal results occur, and remind medical staff to intervene manually; ④ Researchers can view the recent health status of patients through the terminal, and members of corresponding disciplines can give targeted health guidance according to the existing health problems of patients; Remind patients with complex conditions to have outpatient reexamination; ⑤ Push disease related knowledge every week for patients to learn independently.
  Interventions: Device: integrated care mode
- Control group based on conventional care mode (Active Comparator): ① The health education manual for patients receiving targeted treatment of gastric stromal tumors will be issued. The patients who need targeted treatment will be identified and followed up in the routine outpatient department (1 month, 3 months, 6 months, 12 months after surgery, and once a year thereafter); ② Telephone follow-up (1 month, 3 months, 6 months, 12 months and once a year thereafter); ③ Patients independently complete disease symptom monitoring, lifestyle adjustment, and other disease self-management.
  Interventions: Device: conventional care mode

INTERVENTIONS:
Device: integrated care mode — The information system consists of big data platform and nursing strategy platform. The system includes medical work end, patient operation end and administrator management end. The big data platform can automatically extract patient data from HIS, Medcare and other patient diagnosis and treatment systems, complete registration and establish patient health files according to the preset patient registration standards. By comparing the data input on the patient side with the database set on the platform, the system decision-making module can generate personalized measures and plans for feedback to patients, and can generate patient information overview feedback to the nurse side. Complete intelligent push of symptom management decision model
  Arms: Experimental group based on integrated care mode
Device: conventional care mode — ① The health education manual for patients receiving targeted treatment of gastric stromal tumors will be issued. The patients who need targeted treatment will be identified and followed up in the routine outpatient department (1 month, 3 months, 6 months, 12 months after surgery, and once a year thereafter); ② Telephone follow-up (1 month, 3 months, 6 months, 12 months and once a year thereafter); ③ Patients independently complete disease symptom monitoring, lifestyle adjustment, and other disease self-management.
  Arms: Control group based on conventional care mode

SUMMARY:
The goal of this clinical trial is to construct a symptom management strategy for patients with gastrointestinal stromal tumor targeted therapy based on symptom management theory under the guidance of MRC framework. Embed the symptom management strategy into the information platform and conduct an empirical study on integrated care for GIST patients, and compare it with the traditional outpatient follow-up patients to explore the safety and effectiveness of the symptom management strategy and the application effect of the integrated care platform.

DETAILED DESCRIPTION:
The purpose of this clinical trial is to build an information platform for symptom management and integrated care strategy of gastrointestinal stromal tumor targeted treatment patients: the system is composed of big data platform and care strategy platform. The big data platform can automatically extract patient data from HIS, Medcare and other patient diagnosis and treatment systems according to the pre-set patient inclusion criteria, form a health file of gastrointestinal stromal tumor targeted treatment patients, and complete the enrollment. The system will intelligently promote the care strategies of the patients included in the big data platform, promote the two-way communication between doctors and patients, and realize the functions of timed symptom evaluation, symptom management, symptom management result feedback, etc. All patient health data can be customized output through the big data platform. The two platforms complement each other, promote patient self-management, improve the quality of medical follow-up service, reduce the workload of medical personnel, optimize the use of medical resources, and improve the quality of scientific research data. It is not necessary for patients to judge how to take intervention measures, but the system's management center decision-making module will evaluate the symptoms of patients, and then pop up corresponding measures, so that patients can more effectively cope with the discomfort of related symptoms caused by targeted treatment at home, and alleviate the impact on life.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as gastrointestinal stromal tumor and receiving targeted therapy

  * Over 18 years old, with normal communication ability

    * Will use smart phones, or the family members who will use smart phones will live in the meeting

      * Informed consent and voluntary participation in this study.

Exclusion Criteria:

* Patients with psychiatric history or congenital mental retardation

  * The patient or his/her cohabiting family members cannot complete the health status self test, health status assessment and questionnaire under the prompts of the platform.

Criteria for case termination:

* Those who voluntarily put forward termination during the study period and are unwilling to accept follow-up or refuse to fill in the questionnaire

  * Death

    * Lost subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Scoring of quality of life using the cancer treatment function evaluation system | One month after intervention
  Evaluate the quality of life of patients. The scale consists of 27 items: 7 items of physiological status (coded GP1-GP7), 7 items of social/family status (GS1-GS7), 6 items of emotional status (GE1-GE6) and 7 items of functional status (GF1-GF7). Each item adopts a 5-level scoring method. From "not at all" to "very", the score is 0-4, respectively. Among them, GP1-GP7, GE1, and GE3-GE6 are reverse items.
Scoring of quality of life using the cancer treatment function evaluation system | Three month after intervention
  Evaluate the quality of life of patients. The scale consists of 27 items: 7 items of physiological status (coded GP1-GP7), 7 items of social/family status (GS1-GS7), 6 items of emotional status (GE1-GE6) and 7 items of functional status (GF1-GF7). Each item adopts a 5-level scoring method. From "not at all" to "very", the score is 0-4, respectively. Among them, GP1-GP7, GE1, and GE3-GE6 are reverse items.
Scoring of quality of life using the cancer treatment function evaluation system | Six month after intervention
  Evaluate the quality of life of patients. The scale consists of 27 items: 7 items of physiological status (coded GP1-GP7), 7 items of social/family status (GS1-GS7), 6 items of emotional status (GE1-GE6) and 7 items of functional status (GF1-GF7). Each item adopts a 5-level scoring method. From "not at all" to "very", the score is 0-4, respectively. Among them, GP1-GP7, GE1, and GE3-GE6 are reverse items.
Quality of life score of patients assessed by the specific module of gastric cancer of Anderson Symptom Assessment Scale | One month after intervention
  It is widely applicable to cancer patients of different types and treatments. The scale consists of two parts, which measure the severity of 13 core cancer symptoms and "symptom interference", that is, the interference of symptoms to patients and the specific module of gastrointestinal cancer. The severity of 13 core symptoms was evaluated for cancer symptoms, including pain, fatigue, nausea, restless sleep, distress, shortness of breath, amnesia, anorexia, drowsiness, dry mouth, sadness, vomiting and numbness, of which 2 items evaluated sleep problems; Symptom interference assessment The interference degree of the above 13 core symptoms to the six daily life items of general activities, work, emotion, walking, interpersonal relationship and fun of life. Each item is scored from 0 to 10 points, 0-4 points are mild, 5-6 points are moderate, and ≥ 7 points are severe.
Quality of life score of patients assessed by the specific module of gastric cancer of Anderson Symptom Assessment Scale | Three month after intervention
  It is widely applicable to cancer patients of different types and treatments. The scale consists of two parts, which measure the severity of 13 core cancer symptoms and "symptom interference", that is, the interference of symptoms to patients and the specific module of gastrointestinal cancer. The severity of 13 core symptoms was evaluated for cancer symptoms, including pain, fatigue, nausea, restless sleep, distress, shortness of breath, amnesia, anorexia, drowsiness, dry mouth, sadness, vomiting and numbness, of which 2 items evaluated sleep problems; Symptom interference assessment The interference degree of the above 13 core symptoms to the six daily life items of general activities, work, emotion, walking, interpersonal relationship and fun of life. Each item is scored from 0 to 10 points, 0-4 points are mild, 5-6 points are moderate, and ≥ 7 points are severe.
Quality of life score of patients assessed by the specific module of gastric cancer of Anderson Symptom Assessment Scale | Six month after intervention
  It is widely applicable to cancer patients of different types and treatments. The scale consists of two parts, which measure the severity of 13 core cancer symptoms and "symptom interference", that is, the interference of symptoms to patients and the specific module of gastrointestinal cancer. The severity of 13 core symptoms was evaluated for cancer symptoms, including pain, fatigue, nausea, restless sleep, distress, shortness of breath, amnesia, anorexia, drowsiness, dry mouth, sadness, vomiting and numbness, of which 2 items evaluated sleep problems; Symptom interference assessment The interference degree of the above 13 core symptoms to the six daily life items of general activities, work, emotion, walking, interpersonal relationship and fun of life. Each item is scored from 0 to 10 points, 0-4 points are mild, 5-6 points are moderate, and ≥ 7 points are severe.
Anxiety tendency of patients in the past week assessed by self rating anxiety scale | One month after intervention
  It can accurately evaluate the anxiety tendency of patients in the past week. The evaluation method is convenient and highly operable. The evaluation time is short and the content is easy to understand. Cronbach's of SAS α The coefficient is 0.824, including 20 items, with a total score of 100 points. In the entry, "1 minute" means no or very little time, "2 minutes" means a small part of time, and "3 minutes" means a considerable amount of time; "4 points" means most or all of the time, in which items 5, 9, 13, 17 and 19 are scored reversely. The integral part of the original score multiplied by 1.25 is the final standard score. The higher the total score, the more obvious the anxiety symptoms of the patient. The score of normal emotion is below 50, the score of mild anxiety is between 50-59, the score of moderate anxiety is between 60-69, and the score of more than 70 is severe anxiety.
Anxiety tendency of patients in the past week assessed by self rating anxiety scale | Three month after intervention
  It can accurately evaluate the anxiety tendency of patients in the past week. The evaluation method is convenient and highly operable. The evaluation time is short and the content is easy to understand. Cronbach's of SAS α The coefficient is 0.824, including 20 items, with a total score of 100 points. In the entry, "1 minute" means no or very little time, "2 minutes" means a small part of time, and "3 minutes" means a considerable amount of time; "4 points" means most or all of the time, in which items 5, 9, 13, 17 and 19 are scored reversely. The integral part of the original score multiplied by 1.25 is the final standard score. The higher the total score, the more obvious the anxiety symptoms of the patient. The score of normal emotion is below 50, the score of mild anxiety is between 50-59, the score of moderate anxiety is between 60-69, and the score of more than 70 is severe anxiety.
Anxiety tendency of patients in the past week assessed by self rating anxiety scale | Six month after intervention
  It can accurately evaluate the anxiety tendency of patients in the past week. The evaluation method is convenient and highly operable. The evaluation time is short and the content is easy to understand. Cronbach's of SAS α The coefficient is 0.824, including 20 items, with a total score of 100 points. In the entry, "1 minute" means no or very little time, "2 minutes" means a small part of time, and "3 minutes" means a considerable amount of time; "4 points" means most or all of the time, in which items 5, 9, 13, 17 and 19 are scored reversely. The integral part of the original score multiplied by 1.25 is the final standard score. The higher the total score, the more obvious the anxiety symptoms of the patient. The score of normal emotion is below 50, the score of mild anxiety is between 50-59, the score of moderate anxiety is between 60-69, and the score of more than 70 is severe anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Li Chen, Bachelor, Study Chair — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Nanjing Drum Tower Hospital, The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No